CLINICAL TRIAL: NCT00003969
Title: A Phase I Pharmacokinetic and Pharmacodynamic Study of 17-Allylamino-17-Demethoxygeldanamycin (17-AAG) (NSC 330507) Via Intravenous Administration in Patients With Advanced Malignancies
Brief Title: Geldanamycin Analogue in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CRC-PHASE-I-PH1/074; CDR0000067170 (Registry Identifier: PDQ (Physician Data Query)); NCI-T99-0013; EU-99055
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2000-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — tanespimycin

INTERVENTIONS:
Drug: tanespimycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase I trial is studying the side effects and best dose of a geldanamycin analogue in treating patients with advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose for a geldanamycin analogue, 17-allylamino-17-demethoxygeldanamycin (AAG), in patients with advanced malignancies.
* Determine the toxic effects and dose-limiting toxicity of AAG in this patient population.
* Determine the safe dose of AAG for a Phase II study.
* Measure the pharmacokinetic and pharmacodynamic profiles of AAG in these patients.
* Assess time to tumor progression and any antitumor activity in patients treated with AAG.

OUTLINE: This is a dose-escalation study.

Patients receive a geldanamycin analogue, 17-allylamino-17-demethoxygeldanamycin (AAG), IV over 15-30 minutes every week. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of AAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: Approximately 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven malignancies refractory to conventional treatment or for which no standard therapy exists
* Primary brain tumor or brain metastases allowed if stable symptoms within 2 weeks prior to study and able to give informed consent

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* WHO 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL
* Absolute neutrophil count at least 1,500/mm^3

Hepatic:

* Bilirubin less than 1.0 mg/dL
* AST and ALT no greater than 2.5 times upper limit of normal if due to liver metastases
* No chronic liver disease

Renal:

* Creatinine less than 1.47 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No myocardial infarction within the past 6 months
* No angina requiring treatment within the past 6 months
* No uncompensated coronary artery disease by electrocardiogram or physical examination
* No prior transient ischemic attacks, stroke, or peripheral vascular disease
* LVEF at least 45%

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after study
* No allergy to egg products
* No nonmalignant systemic disease that would increase risk
* No active uncontrolled infection
* No diabetes mellitus with evidence of severe peripheral vascular disease or diabetic ulcers

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) and recovered
* No other concurrent chemotherapy

Endocrine therapy:

* At least 4 weeks since other prior endocrine therapy and recovered
* Concurrent corticosteroids for symptom control allowed if no change in dose requirement within 2 weeks prior to study

Radiotherapy:

* At least 4 weeks since prior radiotherapy (except for palliative reasons) and recovered
* Concurrent radiotherapy allowed for control of bone pain or as indicated

Surgery:

* Not specified

Other:

* No other concurrent investigational treatment
* No concurrent treatment with drugs interfering with hepatic CYP3A4 metabolism (e.g., grapefruit juice or warfarin)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-08; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of 17-allylamino-17-demethoxygeldanamycin (17-AAG) at 4 weeks

SECONDARY OUTCOMES:
Heat shock protein 90 (HSP90) client protein and co-chaperone changes during first course of treatment
Pharmacokinetic profile of 17-AAG during the first course of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ian R. Judson, MA, MD, FRCP, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust - London, London, England, United Kingdom

REFERENCES:
- [Result] Banerji U, O'Donnell A, Scurr M, Pacey S, Stapleton S, Asad Y, Simmons L, Maloney A, Raynaud F, Campbell M, Walton M, Lakhani S, Kaye S, Workman P, Judson I. Phase I pharmacokinetic and pharmacodynamic study of 17-allylamino, 17-demethoxygeldanamycin in patients with advanced malignancies. J Clin Oncol. 2005 Jun 20;23(18):4152-61. doi: 10.1200/JCO.2005.00.612. PMID 15961763